CLINICAL TRIAL: NCT04274413
Title: Assessing CFTR Function in Patients With CFTR Related Pancreatitis Using a Novel Sweat Test
Brief Title: CFTR Related Pancreatitis Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to funding and Covid-19 pandemic
Sponsor: The Hospital for Sick Children (Other)
Collaborators: The National Pancreas Foundation (Other)
Responsible Party: Principal Investigator, Tanja Gonska, Associate Professor and Senior Associate Scientist, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1000065960
Record Dates: First submitted 2020-02-16; First posted 2020-02-18 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Cystic Fibrosis; CFTR Gene Dysfunction
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: Evaporimeter TEWL probes, model RG-1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interventional Arm (Experimental): All patients consented to study will undergo study intervention which is Beta-adrenergic sweat test (Beta sweat test) using evaporimeter. It takes about 60 minutes to complete this test. Once this test is completed, patient will be considered to have completed the study.
  Interventions: Combination Product: Beta Adrenergic Sweat Test

INTERVENTIONS:
Combination Product: Beta Adrenergic Sweat Test — In Beta Sweat Test - sweat secretion will be stimulated by injecting a series of drugs within the skin surface. Small needles will be used to inject minute amounts of each drug. Before and after each skin injection, the skin will be cleaned using an alcohol swab.
  1. Two sensor probes will be strapped to the forearm with rubber bands in position just above the injection site.
  2. Under the first probe, injection atropine will be given in one small area of the skin.
  3. Under the second probe, first injection carbachol will be given in one small area of the skin.
  4. Next, at the second probe area, the normal sweating will be stopped for awhile by injecting a drug called atropine.
  5. Lastly, beta-adrenergic sweating will be stimulated by injecting a combination of the following drugs: atropine, isoproterenol, and aminophylline (β-cocktail). Using probes, all sweat rate readings will be recorded.

SUMMARY:
The main causes of acute recurrent pancreatitis (ARP) or chronic pancreatitis (CP) in children are defects in genes that have been associated to pancreatitis. Among these gene defects CFTR gene mutations are commonly found, 34% ARP and 23% CP . Since not every CFTR gene mutations clinically manifest, just identifying these CFTR gene mutations may not help to establish a clear role of this defect in the etiology of the individual ARP/CP. The novel beta-adrenergic sweat secretion test is a very sensitive test to detect small abnormalities in CFTR function in form of a linear gene-function relation. By identifying even mild CFTR defects, in future will help in finding the role of CFTR modulators and providing treatment to these patients.

ELIGIBILITY:
Inclusion Criteria:

* Age : 4 years and older
* Diagnosis: Acute recurrent pancreatitis or chronic pancreatitis
* History: at least one of the following:

  1. Carry one or two CFTR mutations
  2. Borderline sweat chloride levels
  3. Has Family History of CF
  4. Has had positive CF Newborn screening

     Exclusion Criteria:
* Pregnant females: will be excluded at screening.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Assessment of CFTR function using the Beta Adrenergic Sweat Secretion Test | 60 mins
  CFTR function assessment of patients with acute recurrent or chronic pancreatitis by using Beta adrenergic sweat test.